CLINICAL TRIAL: NCT00848848
Title: A Phase Ib, Multi-Center, Randomized, Observer-Blind, Proof of Concept, Dose- and Formulation-Ranging Study to Evaluate Safety, Tolerability, and Immunogenicity of One Dose of Trivalent Inactivated Influenza Vaccine in Different Presentations (Intramuscular and Intradermal Delivery), Dosages (Regular or Higher A/H3N2 Content) and Doses of Adjuvant Administered to Healthy Elderly Aged ≥ 65 Years
Brief Title: Safety, Tolerability, and Immunogenicity of Different Combinations of Trivalent Influenza Vaccine Varying Influenza Antigen Dose, Adjuvant Dose, and Route of Administration in Healthy Elderly Individuals Ages 65 Years and Older
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seqirus (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: V104P3; 2008-002625-36
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Influenza
Keywords: Influenza; Flu; Vaccine; Intradermal; Adjuvant
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant

ARMS (10):
- 1 (Active Comparator)
  Interventions: Biological: Trivalent Influenza Vaccine
- 2 (Active Comparator)
  Interventions: Biological: Trivalent Influenza Vaccine + high A
- 3 (Active Comparator)
  Interventions: Biological: Trivalent Influenza Vaccine + ¼ dose adjuvant
- 4 (Active Comparator)
  Interventions: Biological: Trivalent Influenza Vaccine + high A + ¼ dose adjuvant
- 5 (Active Comparator)
  Interventions: Biological: Trivalent Influenza Vaccine + ½ dose adjuvant
- 6 (Active Comparator)
  Interventions: Biological: Trivalent Influenza Vaccine + high A + ½ dose adjuvant
- 7 (Active Comparator)
  Interventions: Biological: Trivalent Influenza Vaccine + adjuvant
- 8 (Active Comparator)
  Interventions: Biological: Trivalent Influenza Vaccine + high A + adjuvant
- 9 (Active Comparator)
  Interventions: Biological: Trivalent Influenza Vaccine intradermal dose
- 10 (Active Comparator)
  Interventions: Biological: Trivalent Influenza Vaccine + high A intradermal dose

INTERVENTIONS:
Biological: Trivalent Influenza Vaccine — 1 dose of Trivalent Influenza Vaccine
  Arms: 1
Biological: Trivalent Influenza Vaccine + high A — 1 dose of Trivalent Influenza Vaccine with high A content
  Arms: 2
Biological: Trivalent Influenza Vaccine + ¼ dose adjuvant — 1 dose of Trivalent Influenza Vaccine plus ¼ dose adjuvant
  Arms: 3
Biological: Trivalent Influenza Vaccine + high A + ¼ dose adjuvant — 1 dose of Trivalent Influenza Vaccine with high A plus ¼ dose adjuvant
  Arms: 4
Biological: Trivalent Influenza Vaccine + ½ dose adjuvant — 1 dose of Trivalent Influenza Vaccine plus ½ dose adjuvant
  Arms: 5
Biological: Trivalent Influenza Vaccine + high A + ½ dose adjuvant — 1 dose of Trivalent Influenza Vaccine with high A plus ½ dose adjuvant
  Arms: 6
Biological: Trivalent Influenza Vaccine + adjuvant — 1 dose of Trivalent Influenza Vaccine plus adjuvant
  Arms: 7
Biological: Trivalent Influenza Vaccine + high A + adjuvant — 1 dose of Trivalent Influenza Vaccine with high A plus adjuvant
  Arms: 8
Biological: Trivalent Influenza Vaccine intradermal dose — 1 dose of Trivalent Influenza Vaccine intradermal dose
  Arms: 9
Biological: Trivalent Influenza Vaccine + high A intradermal dose — 1 intradermal dose of Trivalent Influenza Vaccine + high A
  Arms: 10

SUMMARY:
The study will evaluate the safety, tolerability and immunogenicity of different doses and types of Influenza Vaccine in healthy elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 65 years or older generally in good health as determined by medical history, physical assessment and clinical judgment of the investigator.

Exclusion Criteria:

* Subjects who have received influenza vaccine within the past 6 month and who have received adjuvanted vaccine in the past two years.
* Subjects with hypersensitivity to vaccine components. Subjects who are on or were recently on immunosuppressive therapy.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 450 (Actual)
Dates: Start 2008-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Assessment of all adverse events from time of vaccination through study end will be collected to for safety assessment. | 21 days

SECONDARY OUTCOMES:
Strain-specific influenza antibody titers will be used to assess Immunogenicity | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- Center For Vaccinology, Ghent, Belgium

REFERENCES:
- [Derived] Della Cioppa G, Nicolay U, Lindert K, Leroux-Roels G, Clement F, Castellino F, Galli C, Groth N, Levin Y, Del Giudice G. A dose-ranging study in older adults to compare the safety and immunogenicity profiles of MF59(R)-adjuvanted and non-adjuvanted seasonal influenza vaccines following intradermal and intramuscular administration. Hum Vaccin Immunother. 2014;10(6):1701-10. doi: 10.4161/hv.28618. Epub 2014 Apr 14. PMID 24732325
- [Derived] Della Cioppa G, Nicolay U, Lindert K, Leroux-Roels G, Clement F, Castellino F, Galli G, Groth N, Del Giudice G. Superior immunogenicity of seasonal influenza vaccines containing full dose of MF59 ((R)) adjuvant: results from a dose-finding clinical trial in older adults. Hum Vaccin Immunother. 2012 Feb;8(2):216-27. doi: 10.4161/hv.18445. Epub 2012 Feb 1. PMID 22426371